CLINICAL TRIAL: NCT02681770
Title: Individual and Dyadic Functioning of Patients and Their Spouses After Kidney Transplantation With Regard to Adherence and Quality of Life
Brief Title: Individual and Dyadic Functioning, Adherence, and Quality of Life After Kidney Transplantation
Acronym: IDyAL
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Weusthoff, Dr. Sarah, post-doctoral research associate, Hannover Medical School
Other Study IDs: 3003-2016
Record Dates: First submitted 2016-02-01; First posted 2016-02-12 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Transplantation; Family Characteristics
Keywords: kidney transplantation; adherence; quality of life; couples; fundamental frequency; communication; social support
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Following solid organ transplantation, adherence to treatment regime (especially with regard to a reliable intake of immunosuppressant medication) is crucial for transplant survival, and has an impact on the patients' health and morbidity. Approximately 35 % of graft rejection or failure cases in kidney transplant patients are due to insufficient levels of adherence or non-adherence to immunosuppressant medication. Adherence is influenced by both individual and interpersonal aspects in complex interaction.

This study aims at investigating individual and dyadic functioning of both patients and their spouses following kidney transplantation. Outcome measures of interest are patient's level of adherence and both patient and spouse's subjective quality of life.

DETAILED DESCRIPTION:
In Germany, kidney transplant patients form the largest group in solid organ transplantation. Improvements in diagnosing and treating medical problems and complications have lead to enhanced survival rates after transplantation. A crucial factor for the long-term success of kidney transplantations is the patients' life-long adherence to immunosuppressant medication. Numerous aspects influencing adherence have been investigated empirically. Across studies, social support has been shown to have an important impact on levels of patients' adherence to treatment. In kidney patients, lower levels of social support have been found to be a risk factor for non-adherence to immunosuppressant therapy, and impaired integration of the transplantation.

From other long-term and potentially life-threatening medical conditions such as breast cancer, the patients' husbands/wives, or spouses are often the primary source of (social) support and of central importance with regard to treatment-related decisions. Thus, spouses are important agents in the course of treatment but are also under considerable (additional) strain. Most studies on psychosocial outcomes of organ transplantation have focused on either patients or spouses. However, medical, social, and psychological aspects influence transplantation outcomes and patients' as well as spouses functioning in complex interaction and should be investigated accordingly.

The study at hand aims at investigating the nature of marital / relationship quality and communication, social support behaviors, emotional arousal, and psychological distress in patients and their spouses after kidney transplantation. Additionally, the role of these variables of interest for important post-transplantation outcomes such as the patients' adherence to immunosuppressive medication and quality of life in both patients and spouses will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplantation six or more months ago
* treated with immunosuppressive medication
* no Episode of acute rejection reported
* in a Long-term relationship (Duration of 12 or more months)
* spouse accompanying Patient to transplantation outpatient clinic

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a kidney transplantation at Hannover Medical School presenting for monthly follow-up appointments at the nephrological transplantation outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
levels of adherence (externally evaluated and self-reported, both via questionnaires) | 6 months after kidney transplantation
  self-reported (by Patient) and externally evaluated (by spouse) adherence to immunosuppressive medication

SECONDARY OUTCOMES:
social support behaviors (self-report questionnaires and coding systems) | 6 months after kidney transplantation
  self-reported and observed communication behavior and self-rated marital quality
emotional functioning (self-report questionnaire and physiological assessment) | 6 months after kidney transplantation
  self-reported and objectively assessed levels of Emotion regulation and emotional arousal in patients and spouses during social Support interactions with each other after kidney transplantation
quality of life (self-report questionnaire) | 6 months after kidney transplantation
  self-reported quality of life in patients and spouses after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Zimmermann, Professor, Study Director — Hannover Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Low JK, Williams A, Manias E, Crawford K. Interventions to improve medication adherence in adult kidney transplant recipients: a systematic review. Nephrol Dial Transplant. 2015 May;30(5):752-61. doi: 10.1093/ndt/gfu204. Epub 2014 Jun 20. PMID 24950938
- [Background] DiMatteo MR. Social support and patient adherence to medical treatment: a meta-analysis. Health Psychol. 2004 Mar;23(2):207-18. doi: 10.1037/0278-6133.23.2.207. PMID 15008666
- [Background] Northouse L, Templin T, Mood D. Couples' adjustment to breast disease during the first year following diagnosis. J Behav Med. 2001 Apr;24(2):115-36. doi: 10.1023/a:1010772913717. PMID 11392915
- [Background] Pabst S, Bertram A, Zimmermann T, Schiffer M, de Zwaan M. Physician reported adherence to immunosuppressants in renal transplant patients: Prevalence, agreement, and correlates. J Psychosom Res. 2015 Nov;79(5):364-71. doi: 10.1016/j.jpsychores.2015.09.001. Epub 2015 Sep 18. PMID 26526310
- [Background] Zimmermann T, Pabst S, Bertram A, Schiffer M, de Zwaan M. Differences in emotional responses in living and deceased donor kidney transplant patients. Clin Kidney J. 2016 Jun;9(3):503-9. doi: 10.1093/ckj/sfw012. Epub 2016 Mar 24. PMID 27274840